CLINICAL TRIAL: NCT07047859
Title: Clinical Investigation of Sympathetic Nerve Width Measurement in Thoracoscopic Sympathectomy
Status: Not yet recruiting | Type: Observational
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Jiang Fan, Professor, Tongji University
Other Study IDs: 20250228033833606
Record Dates: First submitted 2025-06-08; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Thoracoscopic Sympathectomy (ETS)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective, single-center observational study evaluates the clinical utility of intraoperative sympathetic nerve width measurement during thoracoscopic sympathectomy (ETS) for palmar/craniofacial hyperhidrosis (PH/CH) and facial blushing (FF). The study aims to correlate nerve width-measured using a novel Rapid Intraoperative Sympathetic Nerve Width System (RMSNW-OS) (±0.2mm precision)-with surgical outcomes, compensatory sweating rates, patient satisfaction, and 12-month efficacy.

Approximately 1,000 patients (aged 18-55) will undergo standardized ETS at Shanghai First People's Hospital (2025-2029). Objective metrics include thermographic (palmar/forehead temperature), hemodynamic (HR/BP), biochemical (catecholamines), and Doppler flow measurements. Patient-reported outcomes use diagnosis-specific binary questionnaires and the Hyperhidrosis Disease Severity Scale (HDSS).

Statistical analysis will determine if nerve width predicts treatment response. Innovations include RMSNW-OS standardization and a multidimensional assessment framework to optimize ETS precision and patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis : Confirmed autonomic nervous dysfunction (including palmar hyperhidrosis, craniofacial hyperhidrosis, or facial blushing).
2. Age : ≥18 years and ≤55 years.
3. Cardiopulmonary Function :

   Normal preoperative chest CT scan and electrocardiogram (ECG).
4. Performance Status : ECOG score (see Attachment 1) of 0-1, indicating good clinical fitness and ability to perform daily activities independently.
5. Informed Consent : Patients and their families fully understand the study's purpose, procedures, risks, and potential benefits, voluntarily sign the Informed Consent Form, and agree to participate.

Exclusion Criteria:

1. Abnormal Preoperative ECG :

1. Severe arrhythmias:

   1. Type II second-degree or higher atrioventricular block.
   2. Symptomatic ventricular arrhythmias.
   3. Uncontrolled supraventricular arrhythmias (resting heart rate >100 bpm). These may cause inadequate cardiac output, hypoperfusion of vital organs, and increased surgical risk.
2. Myocardial ischemia or infarction:

   1. ECG showing ST-segment elevation/depression, T-wave inversion.
   2. Pathological Q-waves indicating myocardial infarction. 2. Abnormal Chest CT :

1) Severe pulmonary infections (e.g., lobar pneumonia, empyema) with symptoms like fever, cough, dyspnea. Surgery increases infection risk and may lead to atelectasis or respiratory failure.

2) Pneumothorax or tension pneumothorax:

1. Significant lung collapse causing dyspnea.
2. Tension pneumothorax requiring immediate chest tube drainage. 3) Pleural effusion (moderate/large volume): Causes dyspnea or mediastinal shift; surgery may worsen respiratory function.

   3. Hyperthyroidism-induced facial blushing or generalized hyperhidrosis. 4. Anesthesia Contraindications : Allergy to anesthetics or high-risk conditions (severe pulmonary/cardiac dysfunction).

   5. Cognitive/Psychiatric Impairment : Inability to provide informed consent or understand study risks.

   6. Non-Compliance with Follow-up : Inability to adhere to postoperative visits.

   7. Immunodeficiency Disorders : Severe immunodeficiency, AIDS, or organ transplant history.

   8. Frailty/Advanced Age : Elderly patients with comorbidities or functional decline unfit for surgery.

   9. Severe Organ Dysfunction : Cirrhosis, renal failure, or inability to tolerate surgery/recovery.

   10. Active Infections : Under antibiotic treatment for pneumonia, tuberculosis, or bacterial infections.

   11. Uncontrolled Diabetes : Poor glycemic control with complications (retinopathy, diabetic foot).

   12. Concurrent Clinical Trials : Participation in other interventional studies affecting results.

   13. Severe Malnutrition : Significant weight loss or nutritional deficiency increasing anesthesia/surgical risks.

   14. Hematologic Disorders : Anemia, thrombocytopenia, or coagulopathies affecting hemostasis/recovery.

   15. Severe Chronic Respiratory Failure : Long-term ventilator dependence or tracheostomy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Target Cohort : Adults (18-55 years) diagnosed with primary autonomic dysfunction disorders eligible for thoracoscopic sympathectomy (ETS):
  Palmar Hyperhidrosis (PH) : Excessive sweating of the hands. Craniofacial Hyperhidrosis (CH) : Excessive sweating of the head/face. Facial Blushing (FF) : Uncontrolled facial erythema.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative Sympathetic Nerve Width | Intraoperative (Day 0)
  Quantitative measurement (mm) of thoracic sympathetic nerve trunks (T2 for craniofacial hyperhidrosis/facial blushing; T4 for facial blushing), using the Rapid Measurement System (RMSNW-OS). Measurement based on thoracoscopic image pixel ratios. Method: Calibrated electrosurgical hook with 5 mm reference; width calculated from still-frame images. Precision: ±0.2 mm.
Predictive Value of Nerve Width for Surgical Success | through study completion, an average of 1 year
  Assess whether intraoperative sympathetic nerve width (mm) predicts surgical success, defined as ≥50% symptom reduction based on the Hyperhidrosis Disease Severity Scale (HDSS). Analysis Method: ROC curve analysis.
Predictive Value of Nerve Width for Compensatory Hyperhidrosis | through study completion, an average of 1 year
  Assess whether intraoperative sympathetic nerve width (mm) predicts the incidence of clinically significant compensatory hyperhidrosis requiring intervention. Analysis Method: ROC curve analysis.
Symptom Recurrence Rate | 6/12 months post-op vs. 1-month baseline.
  Proportion of patients reporting recurrence of primary symptoms (palmar hyperhidrosis, craniofacial hyperhidrosis, or facial blushing) at follow-up.
Sustained Quality of Life Improvement | 6/12 months post-op vs. 1-month baseline.
  Improvement in patient-reported quality of life scores, measured by validated questionnaires, compared to 1-month postoperative baseline.
Palmar/Forehead Temperature Change | Baseline (pre-op), 1/3/6/12 months post-op.
  ∆ Temperature (°C) pre- vs. post-surgery measured by standardized infrared thermometer. Reflects sympathetic denervation effect on peripheral circulation.
Patient Satisfaction | 1/3/6/12 months post-op.
  Proportion of patients reporting improvement in social confidence, daily functioning, and symptom burden using binary (yes/no) responses from diagnosis-specific questionnaires. Unit of Measure: Percentage of patients responding "Yes"
Hyperhidrosis Disease Severity Scale (HDSS) Score | 1/3/6/12 months post-op.
  Change in HDSS score (scale 1-4) to assess severity of hyperhidrosis and its impact on daily life. Unit of Measure: Units on a 4-point scale.
Compensatory Hyperhidrosis Rate | 1/3/6/12 months post-op.
  Incidence (%) of clinically significant compensatory sweating (patient-reported or physician-confirmed).

SECONDARY OUTCOMES:
Operative Time | Intraoperative (Day 0).
  Duration of surgery measured from skin incision to final skin closure, recorded in minutes.
Intraoperative Blood Loss | Intraoperative (Day 0).
  Volume of blood lost during surgery, measured using suction canister collection and gauze weight difference.
Resting Heart Rate | Baseline (pre-op), 1/3/6/12 months post-op.
  Measurement of resting heart rate (beats per minute) at baseline and postoperatively to assess autonomic function changes. Unit of Measure: Beats per minute (bpm).
Resting Blood Pressure | Baseline (pre-op), 1/3/6/12 months post-op.
  Measurement of systolic and diastolic blood pressure (mmHg) at rest to evaluate hemodynamic changes. Unit of Measure: Millimeters of mercury (mmHg).
Plasma Catecholamine Levels | Baseline (pre-op), 1/3/6/12 months post-op.
  Quantification of dopamine, epinephrine, and norepinephrine levels in plasma.
Blood Flow Velocity | Baseline (pre-op), 1/3/6/12 months post-op.
  Doppler ultrasound-derived flow velocity (cm/s) in hands/forehead:
  Vm (Mean Velocity) = [Peak Systolic (Vs) + 2×End-Diastolic (Vd)] / 3.
Serum Electrolyte Levels | Baseline (pre-op), 1/3/6/12 months post-op.
  Measurement of sodium (Na⁺), potassium (K⁺), and chloride (Cl-) levels in serum to monitor electrolyte balance.
Liver Function Tests | Baseline (pre-op), 1/3/6/12 months post-op.
  Measurement of liver enzymes (ALT, AST) to assess potential organ toxicity.
Kidney Function Tests | Baseline (pre-op), 1/3/6/12 months post-op.
  Measurement of kidney function markers (creatinine, BUN) to assess potential organ toxicity.
White Blood Cell (WBC) Count | Baseline (pre-op), 1/3/6/12 months post-op.
  Measurement of white blood cell count to monitor for infection, inflammation.
Red Blood Cell (RBC) Count | Baseline (pre-op), 1/3/6/12 months post-op.
  Measurement of red blood cell count to assess anemia risk.
Platelet Count | Baseline (pre-op), 1/3/6/12 months post-op.
  Measurement of platelet count to evaluate clotting potential and risk of thrombocytopenia.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Zhou, Doctor, Principal Investigator — Shanghai General Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Hongkou Distri 200080
Locations (1):
- Shanghai General Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided